CLINICAL TRIAL: NCT06961721
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase IV Clinical Trial to Evaluate the Immunogenicity and Safety of a Live Attenuated Herpes Zoster Vaccine in Adults Aged 40 Years and Older
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: Inner Mongolia Center for Disease Control and Prevention (Unknown); Center for Disease Control and Prevention, Fujian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PFDP20241008
Record Dates: First submitted 2025-04-23; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Prevention of Herpes Zoster
Keywords: IV Clinical Trial; Herpes Zoster Vaccine, Live; Herpes Zoster; Prevention of Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental vaccine：Herpes Zoster Vaccine, Live (Experimental): After reconstitution, 0.5 ml per bottle. The dose per person is 0.5 ml.
  Interventions: Biological: Herpes Zoster Vaccine, Live
- Identical to the test vaccine but without the varicella-zoster virus. (Placebo Comparator): After redissolving, 0.5 ml per bottle. The dose is 0.5 ml per dose for human and does not contain varicella-zoster live virus.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Herpes Zoster Vaccine, Live — assigned to the vaccine group and placebo group in a 2:1 ratio.
  Arms: Experimental vaccine：Herpes Zoster Vaccine, Live
Biological: Placebo — assigned to the vaccine group and placebo group in a 2:1 ratio.
  Arms: Identical to the test vaccine but without the varicella-zoster virus.

SUMMARY:
To evaluate the immunogenicity 42 days after vaccination with the live attenuated herpes zoster vaccine.

To evaluate the safety of the live attenuated herpes zoster vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years on enrollment day；
2. The informed consent of the subject can be obtained and signed；
3. The subjects themselves were able to complete the trial in accordance with the requirements of the clinical trial protocol；
4. Armpit body temperature ≤37.0℃ on the day of enrollment.

Exclusion Criteria:

1. People who are immune deficient or immunosuppressed due to certain diseases or treatments. Causes of immunodeficiency or immunosuppression may include, but are not limited to, primary or acquired immunodeficiency conditions, such as AIDS or other diseases caused by viral infection; Leukemia, lymphoma, or other malignancies affecting the bone marrow or lymphatic system; Being treated for immunosuppression; Being treated with radiation/chemotherapy for a tumor；
2. Do not use in persons with a history of allergic reaction to any of the components contained in this product；
3. Those who are in the acute stage of acute infection and chronic infection should postpone the vaccination of this product；
4. Premenopausal women who tested positive for pregnancy, pregnant women, breastfeeding women, or those who planned to have a baby within 6 months；
5. If this product and other injectable live attenuated vaccines are not administered at the same time, the interval should be at least 28 days；
6. Treatment with whole blood, plasma, or immunoglobulin is given within 5 months or 3 weeks prior to vaccination；
7. Received another investigational drug within 1 month prior to receiving the investigational vaccine/placebo, or is participating in another clinical trial, or plans to use it during the study；
8. Taking or about to take salicylate drugs, including aspirin and difluorosalicylic acid；
9. Patients with abnormal blood pressure that cannot be controlled by medication (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg)；
10. Previous vaccinations against chickenpox or shingles (including use of registered products or participation in clinical trials of chickenpox or shingles vaccine)；
11. Any situation that the investigator considers likely to affect the evaluation of the trial。

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity: | Day 0 and Day 42
  Geometric mean titer (GMT)at Day 0 and Day 42.
Immunogenicity: | Day 0 and Day 42
  geometric mean concentration (GMC) at Day 0 and Day 42.
Immunogenicity: | Day 0 and Day 42
  geometric mean fold increase (GMFI)at Day 0 and Day 42
Immunogenicity: | Day 0 and Day 42
  seroconversion/seroresponse rate (4-fold increase) at Day 0 and Day 42.

SECONDARY OUTCOMES:
Adverse Events | 42 days
  1. Incidence, severity, and causality of solicited local，systemic adverse events within 14 days post-vaccination；
  2. The incidence and severity of unsolicited adverse events within 42 days after vaccination and their association with vaccination；
  3. Incidence of Serious Adverse events (SAE) within 42 days after vaccination。

IPD SHARING:
Plan to Share IPD: Undecided